CLINICAL TRIAL: NCT02600468
Title: Outline of Survey on Long-Term Use of ORENCIA® Intravenous Infusion 250mg
Brief Title: Survey on Long-Term Use of ORENCIA® Intravenous Infusion 250mg
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-516
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who use ORENCIA: Patients who use ORENCIA for the approved indications and who at the start of treatment
  Interventions: Drug: Orencia

INTERVENTIONS:
Drug: Orencia

SUMMARY:
The purpose of this study to collect information on the safety, especially serious infections and malignancies, and efficacy of the long-term use of ORENCIA Intravenous Infusion 250mg in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are beginning to receive the treatment with ORENCIA Intravenous Infusion 250mg under the approved indications, dosage, and administration
* Have available HAQ data
* Have available DAS28-ESR or DAS28- CRP data
* Have no past or present history of malignancies
* Are expected to be followed up for 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's survival and development of malignancies after treatment discontinuation
Sampling Method: Non-Probability Sample
Enrollment: 671 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety measured by number of Adverse events and laboratory abnormalities associated with adverse events | 3 years

SECONDARY OUTCOMES:
Efficacy measured by Patient's survival | 3 years
Efficacy measured by development of malignancies after treatment discontinuation | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx